CLINICAL TRIAL: NCT05782257
Title: A Pilot Study to Evaluate the Feasibility of a Zinc-optimized Gluten-free Diet Compared With Supplements to Treat Zinc Deficiency in Celiac Disease
Brief Title: Zinc Deficiency Treatment in Celiac Disease: Supplementation Versus Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Maria Ines Pinto Sanchez, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14999
Record Dates: First submitted 2022-12-29; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Celiac Disease; Nutrient Deficiency
Keywords: Zinc deficiency; Microbiome; Gastrointestinal and extra-intestinal symptoms; Supplementation; Dietary Treatment; Feasibility
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Supplementation (Active Comparator): Those allocated in this arm will be provided with 90 capsules of gluten-free Zn gluconate 25 mg (7 mg of elemental Zn; Jamieson®) and will be instructed to take 1 tablet daily with a meal and at least 2 hrs apart from other medications, and iron or copper supplements
  Interventions: Dietary Supplement: Zinc Supplementation
- Zinc Optimized Diet (Experimental): Instructions provided by a dietitian to establish a target of 11 mg/day (female) and 14 mg /day (male) provided by Zn-rich food sources, adjusted for dietary phytate intake.
  Interventions: Other: Zn-Optimized Diet

INTERVENTIONS:
Dietary Supplement: Zinc Supplementation — Take one 25mg Zn gluconate tablet daily
  Arms: Zinc Supplementation
Other: Zn-Optimized Diet — Consume 11 mg/day of zinc-rich foods for females and 14 mg/day in males.
  Arms: Zinc Optimized Diet

SUMMARY:
Micronutrient deficiencies are common amongst celiac disease (CeD) patients due to consumption of a restrictive and nutritionally unbalanced gluten-free diet (GFD) in addition to slow intestinal villi healing. Preliminary data of 221 patients attending our Celiac Disease Clinic at McMaster University show that 64% of patients on a GFD have nutrient deficiencies with zinc (Zn) deficiency affecting 48% of treated CeD patients. Dietary supplements are prescribed to treat Zn deficiency and it is unclear whether Zn levels can be restored with optimizing Zn in diet. This project will evaluate the the feasibility of dietary therapy to treat Zn deficiency in CeD in comparison to supplementation. Additional objectives of this pilot study, are to assess the efficacy of Zn optimized GFD compared to Zn supplements in 1) normalizing plasma Zn levels and 2) improving CeD gastrointestinal and extra-intestinal symptoms at 3 and 6 month. Subjects will be recruited from McMaster Celiac clinic. This randomized controlled trial aims to recruit 50 CeD participants with two treatment groups; zinc optimized diet (guided by dietitian to achieve target of 11 mg/day for females and 14 mg /day for males) or zinc oral supplementation (25 mg zinc gluconate tablet/day; 7 mg elemental Zn) with a total study a total study period of 6 months and 4 visits. To be included in the study the investigators require celiac diagnosed patients confirmed through CeD serology and duodenal biopsies adhering to a GFD > 6 months and plasma Zn ≤9.3 µmol/L. Questionnaires will be used to assess presentation of symptoms, dietary adherence, quality of life, depression and anxiety. The trial would be considered to be feasible if the enrolment fraction (i.e., number of enrolled patients /number of eligible patients) is 60% or above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CeD based on specific CeD serology (elevated anti-tissue transglutaminase IgA, deaminated gliadin peptides-Immunoglobulin G or anti-endomysial antibodies IgA) and confirmed by duodenal biopsies showing villous atrophy (Marsh 3a or greater);
* Adopting a gluten-free diet for at least 6 months;
* Untreated Zn deficiency (Zn plasma levels ≤9.3 µmol/L)

Exclusion Criteria:

* Are already on a Zn optimized diet;
* Treatment with Zn supplements or multivitamins containing >11 mg of Zn in the last month;
* Prior allergic reaction to Zn supplements;
* Treatment with antibiotics or probiotics supplements in the last 30 days;
* Pregnancy or lactation
* Current infection in the last 30 days;
* Intestinal obstruction, short gut (remnant bowel <180 cm), or any serious illness considered by the investigator that will interfere with the study procedure or results. Data including medication and supplementation will be recorded in case report form and Zn content added to total Zn in the analysis.
* Untreated pancreatic insufficiency (fecal elastase <200).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Compliance of Dietary Therapy | 6 months
  To assess compliance to a zinc-optimized dietary treatment. Dietary compliance is measured through evaluating zinc levels from biweekly participant food diaries.
Compliance of Supplementation Therapy | 6 months
  To assess compliance to zinc supplementation therapy. Supplementation compliance is measured by pill counting.

SECONDARY OUTCOMES:
Change from Baseline in Zinc Plasma Levels at Month 3 | Baseline and Month 3
  Plasma Zinc will be measured through bloodwork. Normal plasma zinc (pZn) levels: 9.4 ≤ pZn ≤ 15 ug/dL. Change = (Month 3 - Baseline)
Change in Zinc Plasma Levels from Month 3 to Month 6 | Month 3 and Month 6
  Plasma Zinc will be measured through bloodwork. Normal plasma zinc (pZn) levels: 9.4 ≤ pZn ≤ 15 ug/dL. Change = (Month 6- Month 3)
Change from Baseline in Celiac Disease Symptoms at Month 3 | Baseline and Month 3
  The Celiac Symptoms Index (CSI) is a validated disease-specific symptom index in adults with celiac disease. Possible total scores range from 16 (no symptoms) to 80 (worst possible symptoms). Higher scores indicate increase in severity of symptoms. Change = (Month 3 - baseline)
Change in Celiac Disease Symptoms from Month 3 to Month 6 | Month 3 and Month 6
  The Celiac Symptoms Index (CSI) is a validated disease-specific symptom index in adults with celiac disease. Higher scores indicate increase in severity of symptoms. Possible total scores range from 16 (no symptoms) to 80 (worst possible symptoms). Change = (Month 6 - Month 3)
Change from Baseline in Extra-Intestinal Symptoms at Month 3 | Baseline and Month 3
  The Visual Analog Scale (VAS) is a validated subjective measure of acute and chronic pain.
  Possible total scores range from 0 (no symptoms) to 100 (very severe symptoms). Higher scores indicate increase in severity of symptoms. Change = (Month 3 - Baseline).
Change in Extra-Intestinal Symptoms from Month 3 to Month 6 | Month 3 and Month 6
  The Visual Analog Scale (VAS) is a validated subjective measure of acute and chronic pain.
  Possible total scores range from 0 (no symptoms) to 100 (very severe symptoms). Higher scores indicate increase in severity of depression and anxiety. Change = (Month 6 - Month 3).
Change from Baseline in Depression and Anxiety Symptoms at Month 3 | Baseline and Month 3
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire assessing patient anxiety and depression. Possible scores range from 0 (normal) to 21 (abnormal). Higher scores indicate increase in severity of depression and anxiety. Change = (Month 3- Baseline).
Change in Depression and Anxiety Symptoms from Month 3 to Month 6 | Month 3 and Month 6
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire assessing patient anxiety and depression. Possible scores range from 0 (normal) to 21 (abnormal). Higher scores indicate increase in severity of depression and anxiety. Change = (Month 6- Month 3).
Change from Baseline in Intestinal Function at Month 3 | Baseline and Month 3
  Intestinal function/mass is measured by citrulline plasma levels. Normal citrulline levels range from 20-50 umol/L. Higher levels indicate increased intestinal function.
Change from Baseline in Intestinal Function from Month 3 to Month 6 | Month 3 and Month 6
  Intestinal function/mass is measured by citrulline plasma levels. Normal citrulline levels range from 20-50 umol/L. Higher levels indicate increased intestinal function.
Number of Adverse Events per Treatment Group | Baseline-Month 6
  Adverse events will be documented from baseline to the end of the study (6 months) in the Zinc supplementation and Zinc optimized diet group.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Canada